CLINICAL TRIAL: NCT03825042
Title: Effect of an Antioxidants Mix on Cognitive Performance and Well Being: The Bacopa, Licopene, Astaxantina, Vitamin B12
Acronym: BLAtwelve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A. Menarini Industrie Farmaceutiche Riunite S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MEIF/17/BAC-COG/001
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Results first posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2019-02

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: 9-weeks double-blind, randomized, placebo-controlled, parallel-arm superiority study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study treatment was assigned through envelopes randomization system: the site was provided with sealed envelopes, numbered in progressive number starting from R-001, containing the treatment kit to be assigned to the subject. The Investigator will open the first available envelope in progressive order. Inside the envelope there will be the kit number of the treatment to be assigned to that subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food supplement (Experimental): A mix of bacopa, lycopene, astaxanthin and vitamin B12 Dosage form: tablets Dosage: 1 tablet/die Duration: 8 weeks
  Interventions: Dietary Supplement: A mix of bioactive natural compounds
- Placebo (Placebo Comparator): Inactive compound Dosage form: tablets Dosage: 1 tablet/die Duration: 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: A mix of bioactive natural compounds — A mix of bacopa, lycopene, astaxanthin and vitamin B12 in oral tablets
  Arms: Food supplement
Dietary Supplement: Placebo — Inactive compound in oral tablets
  Arms: Placebo

SUMMARY:
Nine-weeks double-blind, randomized, placebo-controlled, parallel-arm superiority study.

The aim of this study is to evaluate the influence of a mix of four bioactive compounds - bacopa, lycopene, astaxanthin and vitamin B12 - on cognitive performance, mood state and well-being in subjects aged ≥ 60 years with no evidence of cognitive dysfunction.

The primary objective of the study is to evaluate the changes in Trial Making Test (TMT) scores from baseline (V2) to 8 weeks of treatment (V4), analyzed in the following hierarchical order: TMT-B, TMT-A and TMT B-A.

Secondary objectives of this study are to evaluate changes from baseline (V2) to 8 weeks of treatment (V4) in Verbal Fluency Test (VFT) score, Montreal Cognitive Assessment (MoCA) score, Mini Mental State Examination (MMSE) score, Rey Auditory Verbal Learning Test (AVLT), psychological well-being as assessed by General Health Questionnaire (GHQ-12), mood states as assessed by the Profile of Mood Stated (POMS), sexual satisfaction as evaluated by the New Sexual Satisfaction Scale (NSSS).

Changes of metabolic parameters from baseline (V2) to 4 weeks of treatment (V3) and from baseline (V2) to 8 weeks of treatment (V4) will be also evaluated as secondary objectives (glucose, insulin, Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, uric acid).

Changes of plasma markers of oxidative stress from baseline (V2) to 4 weeks of treatment (V3) and from baseline (V2) to 8 weeks of treatment (V4) will be evaluated as secondary objectives (8-iso-Prostaglandin F2alpha, Plasma malondialdehyde).

Finally the safety and tolerability of the study product will be assessed.

DETAILED DESCRIPTION:
The study has been conducted in 1 Italian clinical site and involved 80 subjects.

Subjects will be randomly allocated to one of the following groups:

* Group I: mix of the four bioactive compounds (bacopa, lycopene, astaxanthin and vitamin B12), once a day for 8 weeks per os;
* Group II: placebo, once a day for 8 weeks per os.

The study is double blind. Neither the study staff at clinical sites (Investigators, nurses, pharmacist) nor the subject was aware of the treatment assigned.

Each participant attended 4 visits over a total period of about 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥60 years.
2. Subjects who provide written Informed Consent to the study.

Exclusion Criteria:

1. Subjects with cognitive dysfunctions or clinically significant coexisting medical conditions (cardiovascular disease, cerebrovascular events, overt dementia defined by MMSE <27 or other neurological disorders, thyroid disorders, or inflammatory diseases)
2. Subjects with a score on the Geriatric Depression Scale (GDS) >11 in order to avoid confounding due to the influence of concomitant depression on the performance on cognitive tests
3. Current smokers
4. Habitual users of antioxidant supplements (including vitamins C and E)
5. Habitual consumers of chocolate or other cocoa products (daily consumption of any amount)
6. Subjects under treatments with medications known to have antioxidant properties (including statins and glitazones) or to interfere with cognitive functions (including benzodiazepines and antidepressants)
7. Subjects with hypersensitivity to any component of the study medications
8. Subjects who are participating in or having participated in another clinical trial within the previous three months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovambattista GD Desideri, Principal Investigator — U.O.C. Geriatria e Lungodegenza - P.O. SS Filippo e Nicola di Avezzano
Locations (1):
- U.O.C. Geriatria e Lungodegenza - P.O. SS Filippo e Nicola di Avezzano, Avezzano, L'Aquila, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period started on January 2018 and terminated on October 2018. A total of 80 subjetcs have been randomization and 78 completed the study. Each subject has been involved in the study for approximately two months. A total of 4 study visits has been performed for each subject.
Pre-assignment Details: Subjects who provided written informed consent have been subjected to the screening assessments. Subjects who met all inclusion criteria and none of the exclusion criteria have been eligible for the study and have proceeded with the randomization visit after 7 days.
  No wash-out or run-in period was used in this study. 8
Groups:
- Food Supplement: A mix of bacopa, lycopene, astaxanthin and vitamin B12 Dosage form: tablets Dosage: 1 tablet per day Duration: 8 weeks
  A mix of bioactive natural compounds: A mix of bacopa, lycopene, astaxanthin and vitamin B12 in oral tablets
- Placebo: Inactive compound Dosage form: tablets Dosage: 1 tablet per day Duration: 8 weeks
  Placebo: Inactive compound in oral tablets
Period: Overall Study
Arm/Group | Food Supplement | Placebo
Started | 40 | 40
Completed | 38 | 40
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Food Supplement | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 39 | 76
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.88 (1.36) | 62.05 (1.55) | 61.96 (1.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 40 | 40 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 40 | 40 | 80
Trial Making Test (TMT) A [Mean (Standard Deviation); unit: seconds] — TMT, which explores visual-conceptual and visual-motor tracking, is a frequently used neuropsychological test because of its sensitivity to brain damage. TMT is administered in two parts: TMT-A and TMT-B.
  Part A is a visual-scanning, timed task where participants are asked to connect with lines 25 circles numbered from 1 to 25 as quickly as possible. The test is terminated after 5 minutes even if not completed.
  seconds | 25.17 (10.53) | 24.20 (7.37) | 24.68 (8.95)
Trial Making Test (TMT) B [Mean (Standard Deviation); unit: seconds] — TMT, which explores visual-conceptual and visual-motor tracking, is a frequently used neuropsychological test because of its sensitivity to brain damage. TMT is administered in two parts: TMT-A and TMT-B.
  In Part B participants are asked to connect circles containing numbers (from 1 to 13) or letters (from A to L) in an alternate numeric/alphabetical order. The test is terminated in every case after 10 minutes even if not completed.
  seconds | 56.97 (25.37) | 54.64 (21.30) | 55.80 (23.33)

OUTCOME MEASURES:

1. Primary Outcome: Change in Trail Making Test (TMT) B Between Baseline and End of Treatment
Description: Change in Trail Making Test (TMT) B scores from baseline (V2) to 8 weeks of treatment (V4).
  The reduction in the number of seconds the patients take to make the test after the study treatment means an improvement in cognitive functions.
Time Frame: 8 weeks - from baseline to end of study
Population: Intention To Treat
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Food Supplement | Placebo
Number analyzed (Participants) | 38 | 40
seconds | -17.63 (18.93) | 3.46 (13.08)
Statistical Analysis 1: Comparison: Food Supplement vs Placebo; Test type: Superiority; p = 0.0000, ANCOVA; Mean Difference (Final Values) = -21.01, 95% CI 2-sided [-26.80 to -15.20]

2. Primary Outcome: Change Trail Making Test (TMT) A Between Baseline and End of Treatment
Description: Change in Trail Making Test (TMT) A scores from baseline (V2) to 8 weeks of treatment (V4).
  The reduction in the number of seconds the patients take to make the test after the study treatment means an improvement in cognitive functions.
Time Frame: 8 weeks - from baseline to end of study
Population: Intention To Treat
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Food Supplement | Placebo
Number analyzed (Participants) | 38 | 40
seconds | -6.86 (10.00) | -0.37 (5.31)
Statistical Analysis 1: Comparison: Food Supplement; Test type: Superiority; p = 0.0000, ANCOVA; Mean Difference (Final Values) = -6.08, 95% CI 2-sided [-8.45 to -3.61]

3. Primary Outcome: Change in Trail Making Test (TMT) B - Trail Making Test (TMT) A Between Baseline and End of Treatment
Description: Change in Trail Making Test (TMT) B score minus Trail Making Test (TMT) A score from baseline (V2) to 8 weeks of treatment (V4).
  The reduction in the number of seconds the patients take to make the test after the study treatment means an improvement in cognitive functions.
Time Frame: 8 weeks - from baseline to end of study
Population: Intention To Treat
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Food Supplement | Placebo
Number analyzed (Participants) | 38 | 40
seconds | -10.46 (16.62) | 3.84 (11.65)
Statistical Analysis 1: Comparison: Food Supplement vs Placebo; Test type: Superiority; p = 0.0000, ANCOVA; Mean Difference (Final Values) = -14.56, 95% CI 2-sided [-20.02 to -9.11]

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Food Supplement | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/40
Other Adverse Events (participants affected / at risk) | 1/40 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Food Supplement (N=40) | Placebo (N=40)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Food Supplement (N=40) | Placebo (N=40)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT03825042/SAP_000.pdf
  • Study Protocol (2017-10-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT03825042/Prot_001.pdf